CLINICAL TRIAL: NCT07139470
Title: An Open-label, Single-arm, Multicenter Phase I/II Study of Sacituzumab Tirumotecan (Sac-TMT) Plus Anlotinib in Previously Treated Metastatic Triple Negative Breast Cancer (mTNBC).
Brief Title: Sacituzumab Tirumotecan Plus Anlotinib for Metastatic Triple Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-IIT-001
Record Dates: First submitted 2025-08-10; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sac-TMT+anlotinib (Experimental): In the Phase I part, BOIN design was used. There were 3 prespecified doses (sac-TMT 4mg/kg Q2W +anlotinib 8mg Q3W, sac-TMT 4mg/kg Q2W +anlotinib10mg Q3W, sac-TMT 4mg/kg Q2W +anlotinib12 mg Q3W). In the Phase II part, the patients will receive sac-TMT patients Q2W +anlotinib RP2D Q3W. The treatment will continue until disease progression, unacceptable toxic effects, withdrawal from the trial, or death, whichever occurred first.
  Interventions: Drug: Sacituzumab Tirumotecan + anlotinib

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan + anlotinib — Phase I part: 3 prespecified doses (sac-TMT 4mg/kg Q2W +anlotinib 8mg Q3W, sac-TMT 4mg/kg Q2W +anlotinib10mg Q3W, sac-TMT 4mg/kg Q2W +anlotinib12 mg Q3W).
  Phase II part: sac-TMT patients Q2W +anlotinib RP2D Q3W.

SUMMARY:
This is an open-label, single-arm, multicenter phase I/II study to evaluate the safety and efficacy of sac-TMT plus anlotinib in previously treated mTNBC. The study is expected to enroll up to 59 eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing informed consent.
* Histologically and/or cytologically confirmed triple-negative breast cancer (TNBC) based on the most recent biopsy or pathological specimen, including:

  1. Definition of human epidermal growth factor receptor 2 (HER2) negative: immunohistochemistry (IHC) of 0 or 1+; if HER is 2+ by IHC, negative HER2 expression must be confirmed by fluorescence in situ hybridization (FISH);
  2. Estrogen and progesterone receptor negative means that less than 1% of the cells express hormone receptors as indicated by IHC.
* Patients with unresectable locally advanced or metastatic triple-negative breast cancer who have received at least one line of standard of care regimens, including:

  1. Any treatment received by the patients regardless of triple-negative state can be included as one of the standard of care regimens;
  2. For neoadjuvant and/or adjuvant chemotherapy, if relapse or disease progression to unresectable locally advanced or metastatic disease occurs during treatment or within 12 months after discontinuation of treatment (at least 2 cycles have been completed), it will be considered as one of the standard of care regimens;
  3. For patients with documented germline BRCA1/BRCA2 mutations, if they have been treated with an approved PARP inhibitor, then the PARP inhibitor can be considered as one prior standard of care regimens required;
  4. Patients must have progressed on or were intolerable to the treatment during or after the last treatment prior to enrollment.
* Newly diagnosed brain metastases at screening must be stable for ≥4 weeks after local treatment (e.g., radiotherapy) with imaging confirmation.
* Patients must have at least one measurable lesion per RECIST v1.1 criteria; those with only skin or bone lesions cannot be included.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* With an expected survival of ≥ 12 weeks.
* Patients must have adequate organ and bone marrow function (no blood transfusion, recombinant human thrombopoietin, or colony stimulating factor therapy has been received within 2 weeks prior to the treatment), which is defined as follows:

  1. Hematology: neutrophil count (NEUT) ≥ 1.5 × 10^9/L; platelets (PLT) ≥ 100 × 10^9/L; hemoglobin ≥ 90g/L;
  2. Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), for patients with liver metastases, ALT and AST must be ≤ 5 × ULN; Albumin ≥ 30g/L; total bilirubin (TBIL) ≤ 1.5 × ULN;
  3. Renal function: creatinine clearance (Ccr) ≥ 50 ml/min;
  4. Coagulation function: international normalized ratio (INR), activated partial thromboplastin time (APTT) and prothrombin time (PT) ≤ 1.5 × ULN.
* Patients of childbearing potential (male or female) must use effective medical contraception from consent until 6 months after the end of the dosing period.
* Patients voluntarily participate in the study, sign the informed consent form, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

* Previously received any of the following treatments (including in the adjuvant or neoadjuvant setting):

  1. TargetedTROP2therapy;
  2. Any drug treatment targeting topoisomeraseI, including antibody-drug conjugates (ADC) therapy;
  3. Anti-angiogenic drugtherapy.
* Patients with multiple factors affecting oral medication.
* Known to have meningeal metastasis, brainstem metastasis, spinal cord metastasis, and/or compression, active central nervous system (CNS) metastasis. Patients with previously treated brain metastases can participate if clinically stable for at least 4 weeks before dosing and do not require corticosteroids or anticonvulsants for at least 14 days. Patients with untreated asymptomatic brain metastases must require investigator approval.
* Within 3 years before administration having other malignancies (except for those cured by local treatment, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, etc.).
* Presence of any of the following cardiovascular diseases or risk factors:

  1. Within 6 months before administration, myocardial infarction, unstable angina, acute or persistent myocardial ischemia, grade 3 or grade 4 heart failure, symptomatic or poorly controlled severe arrhythmias, cerebrovascular accident, transient ischemic attack, and other severe cardiovascular diseases;
  2. History of myocarditis, primary cardiomyopathy, specific cardiomyopathy, and other myocardial diseases;
  3. Within 3 months before administration, any deep vein thrombosis (if stabilized by low molecular weight heparin or similar drugs≥ 2 weeks, enrollment is allowed), peripheral arterial thromboembolism, pulmonary embolism, or other severe thromboembolic events;
  4. Presence of aortic aneurysm, aortic dissection aneurysm, or other major vascular diseases that may be life-threatening or require surgery within 6 months before administration.
* Uncontrollable systemic diseases as judged by the investigator:

  1. Poorly controlled diabetes (fasting blood glucose≥ 10 mmol/L on two consecutive occasions);
  2. Poorly controlled hypertension (systolic blood pressure> 160 mmHg and/or diastolic blood pressure> 100 mmHg);
  3. Presence of clinically symptomatic or requiring repeated drainage of pleural effusion, pericardial effusion, or ascites (> 1 time/week).
* Presence of steroid-requiring (non-infectious) interstitial lung disease (ILD) or a history of non-infectious pneumonia, currently having ILD or non-infectious pneumonia, or suspected ILD or non-infectious pneumonia that cannot be ruled out by imaging at screening.
* Clinically significant lung damage due to pulmonary complications, including but not limited to any underlying lung disease or any autoimmune, connective tissue, or inflammatory disease that may involve the lungs, or previous total pneumonectomy.
* Patients with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcers, gastrointestinal perforation, abdominal abscess, or acute gastrointestinal bleeding.
* Patients with acute gastrointestinal bleeding, persistent bleeding disorders, or bleeding tendencies such as coagulopathy.
* Toxicity from previous anti-tumor treatments has not recovered to ≤ 1grade (based on NCI CTCAE v5.0 assessment) or to the level specified by the inclusion criteria (excluding toxicities such as alopecia, fatigue, etc., judged by the investigator to be of low safety risk).
* Having an active autoimmune disease requiring systemic treatment in the past two years (including but not limited to: autoimmune hepatitis, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, etc.), systemic treatment includes disease-modifying drugs, immunosuppressants, systemic corticosteroids (> 10 mg/day prednisone or equivalent). Hormone replacement therapy, such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a systemic treatment; within2weeks before administration> 10 mg/day prednisone systemic corticosteroid treatment or other immunosuppressive drugs.
* Known active tuberculosis.
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* With ≥ 2 grade peripheral neuropathy.
* Active hepatitis B or hepatitis C.
* Human Immunodeficiency Virus (HIV) test positive or history of Acquired Immunodeficiency Syndrome (AIDS); known active syphilis infection.
* Known allergy to the study drug or any of its components, known history of severe hypersensitivity to other biological products.
* Major surgery within 4 weeks prior to dosing or expected to require major surgery during the study period.
* Severe infection within 4 weeks prior to dosing, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective treatment within 2 weeks prior to dosing.
* Documented severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or history of corneal disease that impedes delayed corneal healing.
* Non-specific immunomodulatory treatment within 2 weeks prior to dosing (including but not limited to interferon,IL-2), approved traditional Chinese medicine preparations for anti-tumor indications, etc.
* Prior to dosing 30 days after receiving a live vaccine, or planning to receive a live vaccine during the study period.
* Rapid deterioration of the condition during the screening before administration, such as significant changes in physical status.
* Pregnant or breastfeeding women.
* Suffering from local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors, which may lead to high medical risk and/or uncertainty in survival evaluation, such as tumor leukemic reactions, cachexia manifestations, etc.
* Any condition that the researcher believes interferes with the evaluation of the study drug or the safety of the subject or the interpretation of the study results, or any other condition that the investigator believes is not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 60 months
  The primary endpoint of Phase I. ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
  Radiographic assessment of tumor response will be performed based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1
Safety and the recommended phase 2 dose (RP2D) | Up to Day 21
  The primary endpoint of Phase II. BOIN design was used to evaluate the safety and the recommended phase 2 dose (RP2D) of sac-TMT plus anlotinib

SECONDARY OUTCOMES:
Disease control response (DCR) | up to approximately 60 months.
  DCR is defined as the proportion of participants who achieve a complete response (CR) ,partial response (PR) or stable disease (SD).
  Radiographic assessment of tumor response will be performed based on RECIST v1.1
Duration of response (DOR) | up to approximately 60 months
Progression-free survival (PFS) | up to approximately 60 months
Overall Survival (OS) | Until death, up to approximately 60 months.
Health-related quality of life (HRQoL) evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale | up to approximately 60 months
Health-related quality of life (HRQoL) evaluated using the NCC-BC-A scale | up to approximately 60 months
Incidence and severity of adverse events (AEs) | up to approximately 60 months

OTHER OUTCOMES:
Clinical benefit according to TROP2 expression at baseline. | up to approximately 60 months
Clinical benefit according to homologous recombination deficiency (HRD) at baseline | up to approximately 60 months
Clinical benefit according to angiogenesis gene profiles at baseline | up to approximately 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China